CLINICAL TRIAL: NCT03877198
Title: A Randomized Cross-over Trial in the Effect of Automated Oxygen Control Devices on the Distribution of Oxygen Saturation in Preterm Infants
Brief Title: Comparison of Oxygen Controllers in Preterm InfanTs
Acronym: COCkPIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As a result of a slower inclusion rate than expected, competence of medical staff to work with the AVEA ventilator could no longer be guaranteed.
Sponsor: Leiden University Medical Center (Other)
Collaborators: University of Tasmania (Other)
Responsible Party: Principal Investigator, PasABte, Clinical Professor in Pediatrics, Leiden University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: COCkPIT; NL66058.000.18 (Other: Dutch Central Committee on Research Involving Human Subjects)
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Premature Infant; Respiratory Insufficiency; Hypoxia; Hyperoxia
MeSH Terms: conditions — Premature Birth; Respiratory Insufficiency; Hypoxia; Hyperoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor/investigator will be blinded for treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLiO2 (Experimental): Automated oxygen control by the CLiO2 algorithm
  Interventions: Device: Automated oxygen control by the CLiO2 algorithm
- Oxygenie (Experimental): Automated oxygen control by the Oxygenie algorithm
  Interventions: Device: Automated oxygen control by the Oxygenie algorithm

INTERVENTIONS:
Device: Automated oxygen control by the CLiO2 algorithm — Automated oxygen control for 24 hours by the CLiO2 algorithm, preceded by a 1 hour wash-out period
  Other Names: AVEA CLiO2
  Arms: CLiO2
Device: Automated oxygen control by the Oxygenie algorithm — Automated oxygen control for 24 hours by the Oxygenie algorithm, in case of switch in ventilator preceded by a 1-hour wash-out period.
  Other Names: SLE Oxygenie
  Arms: Oxygenie

SUMMARY:
Premature infants often receive respiratory support and supplemental oxygen for a prolonged period of time during their admission in the NICU. While maintaining the oxygen saturation within a narrow target range is important to prevent morbidity, manual oxygen titration can be very challenging. Automatic titration by a controller has been proven to be more effective. However, to date the performance of different controllers has not been compared. The proposed randomized crossover trial Comparing Oxygen Controllers in Preterm InfanTs (COCkPIT) is designed to compare the effect on time spent within target range. The results of this trial will help determining which algorithm is most successful in controlling oxygen, improve future developments in automated oxygen control and ultimately reduce the morbidity associated with hypoxemia and hyperoxemia.

DETAILED DESCRIPTION:
Both hypoxemia as hyperoxemia can potentially be harmful to premature infants. Oxygen titration during respiratory support is vital to prevent these conditions but is very challenging. In the investigator's neonatal intensive care unit preterm infants routinely receive automatic oxygen titration performed by a controller. The currently used controllers are both proven to be more effective than manual titration, however which of the two controllers is most effective in keeping oxygen saturation within target range remains unclear.

This randomized crossover trial tests tests both controllers within every study patient to determine which controller is most effective and thereby would hopefully reduce morbidity associated with hypoxemia and hyperoxemia the most. The primary outcome measure is the proportion of time spent within target range, each controller will be tested for 24 hours within the same study subject. This is excluding a 1-hour wash-out period after a change in ventilator.

Eligible infants are randomized to start with either the Oxygenie algorithm or CLiO2 algorithm and will switch to the other study arm after 24 hours of measurement.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with a gestational age (GA) at birth of 24 - 29+6/7 weeks
* Receiving invasive mechanical ventilation or non-invasive respiratory support (NCPAP or NIPPV)
* Receiving supplemental oxygen (defined as FiO2 ≥ 0.25) at the time of enrollment and for at least 18 hours during the previous 24 hours; Or a coefficient of variation in supplemental oxygen of ≥ 0.1 in the previous 24 hours.
* Expected to complete the 49-hour or 50-hour study period in the current form of respiratory support, i.e. invasive mechanical ventilation or non-invasive respiratory support
* Written informed parental consent must be present.

Exclusion Criteria:

* Major congenital anomalies
* Arterial hypotension requiring vasopressor therapy within 48 hours prior to enrollment.
* If the attending physician considers the infant not stable enough for a switch to another ventilator.

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Proportion of time with SpO2 spent within set target range | Continuously from randomization until study completion. (maximum of 50 hours) Measurements during wash-out periods (up to 1 hour after ventilator switch) will be excluded.
  Total time SpO2 is within the set target range (91-95%) including time spent above target range when in room air (set FiO2 < 0.22)

SECONDARY OUTCOMES:
Proportion of time with SpO2 spent above target range (SpO2 > 95%) | Continuously from randomization until study completion. (maximum of 50 hours) Measurements during wash-out periods (up to 1 hour after ventilator switch) will be excluded.
Proportion of time with SpO2 spent below target range (SpO2 < 91%) | Continuously from randomization until study completion. (maximum of 50 hours) Measurements during wash-out periods (up to 1 hour after ventilator switch) will be excluded.
Coefficient of SpO2 variation | Continuously from randomization until study completion. (maximum of 50 hours) Measurements during wash-out periods (up to 1 hour after ventilator switch) will be excluded.
Time in hypoxemic SpO2 ranges | Continuously from randomization until study completion. (maximum of 50 hours) Measurements during wash-out periods (up to 1 hour after ventilator switch) will be excluded.
  Time in SpO2 range 85-90%, 80-84% and <80%
Time in hyperoxemic SpO2 ranges | Continuously from randomization until study completion. (maximum of 50 hours) Measurements during wash-out periods (up to 1 hour after ventilator switch) will be excluded.
  Time in SpO2 range 96-98% and >98%
Frequency of episodes of hypoxemia | Continuously from randomization until study completion. (maximum of 50 hours) Measurements during wash-out periods (up to 1 hour after ventilator switch) will be excluded.
  Episodes in hypoxemia with SpO2 < 85% for ≥ 30 seconds, for ≥ 60 seconds and hypoxemia < 80% for ≥ 30 seconds and ≥ 60 seconds
Frequency of episodes of hyperoxemia | Continuously from randomization until study completion. (maximum of 50 hours) Measurements during wash-out periods (up to 1 hour after ventilator switch) will be excluded.
  Episodes in hyperoxemia with SpO2 ≥ 97% for ≥ 30 seconds, for ≥ 60 seconds and hyperoxemia ≥ 99% for ≥ 30 seconds and ≥ 60 seconds
Frequency of episodes of bradycardia | Continuously from randomization until study completion. (maximum of 50 hours) Measurements during wash-out periods (up to 1 hour after ventilator switch) will be excluded.
  Episodes where the heart rate < 100 beats per minute for ≥ 10 seconds
Frequency of FiO2 adjustments during automated control | Continuously from randomization until study completion. (maximum of 50 hours) Measurements during wash-out periods (up to 1 hour after ventilator switch) will be excluded.
  FiO2 adjustments as made by the controller and by bedside staff as manual over-rides by the bedside staff as well
Average oxygen exposure | Continuously from randomization until study completion. (maximum of 50 hours) Measurements during wash-out periods (up to 1 hour after ventilator switch) will be excluded.
Coefficient of variation of FiO2 | Continuously from randomization until study completion. (maximum of 50 hours) Measurements during wash-out periods (up to 1 hour after ventilator switch) will be excluded.
Effects on nursing workload in relation to FiO2 adjustment | From randomization until study completion. (maximum of 50 hours) Manual adjustments during wash-out periods will be excluded.
  Number of manual FiO2 adjustments and as the effect on workload measured by a translated questionnaire adapted from the NASA TLX questionnaire, using a visual rating scale
Confidence of the bedside staff in the automated control system | From randomization until study completion. (maximum of 50 hours)
  Measured at the end of each nursing shift by a subset of questions out of the System Trust Scale (Jian et al. 2000) questionnaire. All questions are answered on a 1 (not at all) to 7 (extremely) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Arjan B te Pas, Prof, Principal Investigator — Leiden University Medical Center; Peter A Dargaville, Prof, Principal Investigator — University of Tasmania
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Salverda HH, Cramer SJE, Witlox RSGM, Gale TJ, Dargaville PA, Pauws SC, Te Pas AB. Comparison of two devices for automated oxygen control in preterm infants: a randomised crossover trial. Arch Dis Child Fetal Neonatal Ed. 2022 Jan;107(1):20-25. doi: 10.1136/archdischild-2020-321387. Epub 2021 Jun 10. PMID 34112721